CLINICAL TRIAL: NCT00421031
Title: A Double-Blind, Randomized, Placebo-Controlled Efficacy and Safety Study of DVS-233 SR For Relief of Vasomotor Symptoms Associated With Menopause
Brief Title: Study Evaluating the Safety & Efficacy of DVS-223 SR for Relief of Vasomotor Symptoms Associated With Menopause
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3151A2-315
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Vasomotor Symptoms

INTERVENTIONS:
Drug: DVS-233 SR

SUMMARY:
The purpose of this study is to assess the efficacy and safety of 4 doses of desvenlafaxine-233 sustained release (DVS-233 SR) as compared to placebo for the treatment of moderate to severe vasomotor symptoms associated with menopause, as well as its influence on sleep parameters and other health outcomes indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy, postmenopausal women; at least 12 months of spontaneous amenorrhea or at least 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or at least 6 weeks postsurgical bilateral oophorectomy (with or without hysterectomy).
2. Minimum of 7 moderate to severe hot flushes per day or 50 moderate to severe hot flushes per week at screening:

   * Moderate hot flush: warm sensation with sweating, does not disrupt activity.
   * Severe hot flush: hot sensation with sweating, disrupts activity.
3. Subjects must have body mass index (BMI) less than or equal to 40 using the nomograph for BMI.

Exclusion Criteria:

1. Hypersensitivity to venlafaxine (Effexor or Effexor XR).
2. Use of oral estrogen-, progestin-, androgen-, or SERM-containing drug products within 8 weeks prior to screening; use of transdermal hormone products within 8 weeks prior to screening; use of vaginal hormone products (rings, creams, gels) within 4 weeks prior to screening; use of intrauterine progestins within 8 weeks prior to screening; use of progestin implants or estrogen injectables within 3 months prior to screening; use of estrogen pellet or progestin injectables within 6 months prior to screening.
3. History of a seizure disorder other than a single childhood febrile seizure.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 540
Dates: Start 2003-12; Study Completion 2004-04

PRIMARY OUTCOMES:
The primary objective is to assess the efficacy and safety of 4 doses of DVS-233 SR as compared to placebo for the treatment of moderate to severe VMS associated with menopause.

SECONDARY OUTCOMES:
The secondary objectives are to assess the effects of DVS-233 SR as compared to placebo on sleep parameters and on health outcomes indicators

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (39):
- United States (39):
  - Montgomery, Alabama
  - Peoria, Arizona
  - San Diego, California
  - Stanford, California
  - Colorado Springs, Colorado
  - Newark, Delaware
  - Aventura, Florida
  - Fort Myers, Florida
  - Inverness, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Orange City, Florida
  - Pinellas Park, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - West Venice, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Newburgh, Indiana
  - Lexington, Kentucky
  - Shreveport, Louisiana
  - Portland, Maine
  - Chaska, Minnesota
  - Jackson, Mississippi
  - St Louis, Missouri
  - Billings, Montana
  - Las Vegas, Nevada
  - Reno, Nevada
  - Albuquerque, New Mexico
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Portland, Oregon
  - Erie, Pennsylvania
  - Wexford, Pennsylvania
  - Greenville, South Carolina
  - San Antonio, Texas
  - Norfolk, Virginia

REFERENCES:
- [Derived] Speroff L, Gass M, Constantine G, Olivier S; Study 315 Investigators. Efficacy and tolerability of desvenlafaxine succinate treatment for menopausal vasomotor symptoms: a randomized controlled trial. Obstet Gynecol. 2008 Jan;111(1):77-87. doi: 10.1097/01.AOG.0000297371.89129.b3. PMID 18165395